CLINICAL TRIAL: NCT03791892
Title: The Effects of Shoulder Mobilization Following Supra Scapular Nerve Block in Adhesive
Brief Title: Shoulder Mobilization Following Supra Scapular Nerve Block in Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RiphahI Wajeeha
Record Dates: First submitted 2018-12-31; First posted 2019-01-03 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive capsulitis; suprascapular nerve; shoulder mobilization
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: Experimental
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shoulder mobilization Group (Experimental): Kaltenborn mobilization will be applied to patient in experimental group only.
  Interventions: Other: Shoulder mobilization Group
- Conventional treatment Group (Active Comparator): Application of conventional treatment that includes stretching and strengthening exercises of shoulder.
  Interventions: Other: Conventional Treatment Group

INTERVENTIONS:
Other: Shoulder mobilization Group — Suprascapular nerve block administered every week to both groups. Joint mobilization (3 sets / 40 seconds hold / 30 seconds interval) Stretching exercises (3 sets / 30 seconds hold / 10 seconds interval) Strengthening exercises ( 3 sets / 15 reps)
  Arms: Shoulder mobilization Group
Other: Conventional Treatment Group — Suprascapular nerve block administered every week to both groups. Daily Stretching exercises (3 sets / 30 seconds hold / 10 seconds interval) Daily Strengthening exercises ( 3 sets / 15 reps)
  Arms: Conventional treatment Group

SUMMARY:
Those shoulder patients who fulfill inclusion criteria are divided into two groups. Supervised exercises will be performed by both groups. Kaltenborn mobilization will be applied to patient in experimental group only. Assessment will be done on baseline, 7th and post visit. A total 38 subjects were included in study who met inclusion criteria. Number of patients in both groups was 19.

DETAILED DESCRIPTION:
Adhesive capsulitis is one of the most common debilitating musculoskeletal complaints seen in physiotherapy practice. Adhesive capsulitis is a benign, self-limiting condition of unknown etiology characterized by painful and limited active and passive gleno-humeral range of motion of ≥ 25% in at least two directions most notably shoulder abduction and external rotation. Prevalence of adhesive capsulitis is 2% - 5% in general population.1 Primary adhesive capsulitis and frozen shoulder are current terms used to describe an insidious onset of painful stiffness of the gleno-humeral joint. Secondary adhesive capsulitis, on the other hand, is associated with a known predisposing condition of the shoulder (eg, humerus fracture, shoulder dislocation, avascular necrosis, osteoarthritis, or stroke.

The range of motion (ROM) impairments associated with primary adhesive capsulitis can impact a patient's ability to participate in self-care and occupational activities. Even though this condition is considered self-limiting, with most patients having spontaneous resolution within 3 years, some patients can suffer long-term pain and restricted shoulder motion well beyond 3 years. A disability of this duration places severe emotional and economic hardship on the afflicted person. Most patients are unwilling to suffer this pain, prolonged disability, and sleep deprivation without seeking treatment.

Currently, no standard medical, surgical, or therapy regimen is universally accepted as the most efficacious treatment for restoring motion in patients with shoulder adhesive capsulitis. While physical therapy is commonly prescribed for this condition, some studies have found little treatment benefit. Rehabilitation programs consisting of exercise, massage, and modalities have been shown to improve shoulder ROM in all planes except external and internal rotation. There is evidence, however, that joint mobilization procedures can lessen the associated gleno-humeral rotational deficits characteristic of this condition, especially external rotation. The optimal direction of force and movement application for the joint mobilization to restore external rotation, however, is not clear. Traditionally, physical therapists have used an anterior glide of the humeral head on the glenoid technique to improve external rotation ROM, a choice based on the "convex-on-concave" concept of joint surface motion. In contrast, Roubal et al used a posteriorly directed glide manipulation based on the "capsular constraint mechanism" to restore external as well as internal rotation ROM.Supra-scapular nerve block (SSNB) is a safe and effective method to treat pain in chronic diseases that affect the shoulder. The technique consists of injecting anaesthetics in supraspinatus fossa of affected shoulder, with the patient sitting down and upper limbs pending beside the body.The technique consists of injecting anesthetic in supraspinatus fossa of affected shoulder, with the patient sitting down and upper limbs pending beside the body.3 In this study keltenborn joint mobilization will be use as intervention is to restore the joint play and in order to normalize the rolling and gliding of any joint, which are necessary for the active normal and non-painful movement. Some general exercises also help us to treat adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 70 years
* Both male and female
* Unilateral cases.
* Grade 1 and 2 phase of adhesive shoulder

Exclusion Criteria:

Traumatic /fracture in upper extremity

* Patients with malignancy
* Post-operative shoulder
* Patient under steroid therapy
* Bilateral cases.
* Grade 3 stage of frozen shoulder.
* Patient with sever osteo-arthritis
* Patient with diabetes

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | change from baseline.This tool is used to measure pain intensity
  NPRS) is a scale used to find the level of pain intensity. At the time of treatment session intensity of pain is mainly the center of attention of the treatment. This pain scale is used in routine in clinical setting during the application of treatment procedure to evaluate the intensity of pain. NPRS has good validity and reliability. In our study we evaluate the status of pain in shoulder in individuals with adhesive capsulitis. The NPRS is a segmented numeric version of the visual analog scale in which a respondent selects the whole number (0-10). '0' indicates no pain whereas '10' indicates extreme pain. In our study NPRS values are taken at base line, 7th visit and post visit
Goniometer | change from baseline.This tool is used to measure shoulder ranges
  In physical therapy goniometer is utilized to measures range of movement joint angles in the body.

SECONDARY OUTCOMES:
SHOULDER PAIN AND DISABILITY INDEX (SPADI) | change from baseline.This tool is used to measure shoulder disability
  By using this tool we can access pain as well as level of disability of patient having frozen shoulder. This tool consists of 13 questions. A therapist asked questions to patients. It takes 5 to 10 minutes to finish the questionnaire n marked accordingly. SPADI values were taken at baseline, 7th visit and post visit

CONTACTS AND LOCATIONS:
Overall Officials: imran Amjad, phd*, Principal Investigator — Associate Professor
Locations (2):
- Pakistan (2):
  - Imran Amjad, Islamabad, Punjab Province
  - Riphah International University, Islamabad

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tighe CB, Oakley WS Jr. The prevalence of a diabetic condition and adhesive capsulitis of the shoulder. South Med J. 2008 Jun;101(6):591-5. doi: 10.1097/SMJ.0b013e3181705d39. PMID 18475240
- [Background] Mitchell C, Adebajo A, Hay E, Carr A. Shoulder pain: diagnosis and management in primary care. BMJ. 2005 Nov 12;331(7525):1124-8. doi: 10.1136/bmj.331.7525.1124. No abstract available. PMID 16282408
- [Background] Cho CH, Song KS, Kim BS, Kim DH, Lho YM. Biological Aspect of Pathophysiology for Frozen Shoulder. Biomed Res Int. 2018 May 24;2018:7274517. doi: 10.1155/2018/7274517. eCollection 2018. PMID 29992159
- [Background] Neviaser AS, Hannafin JA. Adhesive capsulitis: a review of current treatment. Am J Sports Med. 2010 Nov;38(11):2346-56. doi: 10.1177/0363546509348048. Epub 2010 Jan 28. PMID 20110457
- [Background] Siegel LB, Cohen NJ, Gall EP. Adhesive capsulitis: a sticky issue. Am Fam Physician. 1999 Apr 1;59(7):1843-52. PMID 10208704
- [Background] Dias R, Cutts S, Massoud S. Frozen shoulder. BMJ. 2005 Dec 17;331(7530):1453-6. doi: 10.1136/bmj.331.7530.1453. PMID 16356983
- [Background] Baums MH, Spahn G, Nozaki M, Steckel H, Schultz W, Klinger HM. Functional outcome and general health status in patients after arthroscopic release in adhesive capsulitis. Knee Surg Sports Traumatol Arthrosc. 2007 May;15(5):638-44. doi: 10.1007/s00167-006-0203-x. Epub 2006 Oct 10. PMID 17031613